CLINICAL TRIAL: NCT01234467
Title: A Phase II Trial of Bendamustine in Combination With Rituximab in Older Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: Bendamustine + Rituximab in Older Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1011; 10-1405 (Other: Office of Human Research Ethics)
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Large B-Cell Lymphoma; Lymphoma, Diffuse Large-Cell; Diffuse Large-Cell Lymphoma; Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Elderly; Newly Diagnosed; Lineberger Comprehensive Cancer Center; University of North Carolina; Bendamustine; Rituximab; Rituxan; Treanda; Phase 2; Geriatric; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine, Rituximab (Experimental): This is a single arm intervention where patients will receive bendamustine at a dose of 120 mg/m^2 infused over 60 minutes in days 1 and 2 of each 21 day cycle along with rituximab 375 mg/m^2 after bendamustine on day 1 of each cycle. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 3 at baseline were allowed to receive bendamustine at a dose of 90 mg/m^2 daily with a dose increase to 120 mg/m^2 daily if their ECOG improved.
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Dosage Form: Intravenous (60 minute infusion) Dosage: 120mg/m2 (ECOG = 0-2) or 90mg/m2 (ECOG = 3) Frequency: Day 1 and Day 2; Every 3 weeks of a 21 day cycle. Duration: 3-6 Cycles
  Other Names: TREANDA; BENDAMUSTINE HYDROCHLORIDE; (NDA) 022249
Drug: Rituximab — Dosage form: Intravenous Dosage: 375 mg/m2 Frequency: Day 1 of every 3 weeks of a 21 day Cycle Duration: 3-6 Cycles
  Other Names: Rituxan; (BLA) 103705

SUMMARY:
The purpose of this research study is to learn about the safety of the treatment with a combination of bendamustine and rituximab and to find out what effects, both good and bad this treatment has on DLBCL. In addition to learning about the combination of bendamustine and rituximab, the researchers are interested in learning about how this cancer treatment affects daily activities. Subjects will be asked to complete a Geriatric Assessment (GA). GAs are designed to gather information on memory, nutritional status, mental health, and level of social support. GAs are also designed to help the health care team understand how well subjects can carry out their day to day activities and to briefly describe what other medical conditions subjects may have. This assessment will help the health care team understand a subject's "functional age" (the age a subject functions at) as compared to a subject's actual age.

The researchers also want to learn how chemotherapy affects the aging process in our bodies. This is done by measuring the amount of p16 in blood. Researchers want to understand if chemotherapy changes the levels of p16 in blood.

DETAILED DESCRIPTION:
This multicenter Phase II clinical study will investigate the complete response (CR) rate after therapy with bendamustine combined with rituximab in older (≥65 years old) patients with previously untreated stage II-IV DLBCL deemed poor candidates for cyclophosphamide, doxorubicin hydrochloride, vincristine (Oncovin®), prednisone, rituximab (CHOP-R); n=37. The hypothesis being tested is that this regimen will be safe and effective as frontline therapy in older DLBCL patients deemed poor candidates for CHOP-R. After 3 cycles of therapy, patients with less than a partial response (PR) will come off study, and be managed at the discretion of their treating physician. Patients who achieve a PR after 3 cycles will continue for a total of 8 cycles of therapy, while patients who achieve a CR will continue for a total of 6 cycles of therapy. Secondary objectives include overall response rates (ORR), disease-free, progression-free and overall survival, and an evaluation of the toxicity and tolerability of the regimen.

This trial also includes an exploratory analysis designed to evaluate a potential correlation between expression of the senescence marker p16INK4a and the toxicity associated with this regimen.

In addition, patients will be asked to participate in a Geriatric Assessment (GA) tool during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated , histologically confirmed, diffuse large B-cell lymphoma (DLBCL), immunophenotyped for CD20
* Age greater than or equal to 65 years
* Stage II-IV
* Measurable disease including lesions that can be accurately measured in 2 dimensions by CT and have a greatest transverse diameter of 1cm or greater, and/or by bone marrow histopathology.
* ECOG performance status of 0-3
* Deemed poor candidate for CHOP-R due to ejection fraction less than or equal to 45%, ECOG performance status of 2, or in the opinion of the treating physician, patient would not tolerate administration of CHOP-R chemotherapy for other reasons,
* Life expectancy of at least 3 months;
* Documented negative serologic testing for HIV, Hepatitis B (unless positive due to prior vaccination), and hepatitis C within the year prior to enrollment
* Adequate bone marrow function (without transfusion support within one week of screening) function:
* Hemoglobin > 8 g/dL
* Absolute neutrophil count (ANC) >1000 cells/mm3
* Platelet count > 75,000/mm3
* Adequate hepatic and renal function as demonstrated by:
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)
* Total serum bilirubin < 2.5 x ULN
* Serum creatinine < 1.5 x ULN
* If sexually active male of reproductive capability, has agreed to use a medically accepted form of contraception from time of enrollment to completion of all follow-up study visits
* Signed an institutional review board (IRB) approved informed consent document

Exclusion Criteria:

* Central nervous system involvement by lymphoma
* History of previous allergic reactions to compounds of similar biological or chemical composition as rituximab or bendamustine
* Medical or other condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective.
* Other active malignancies (except: non-melanoma skin cancer, cervical carcinoma in situ without evidence of disease, prostatic intraepithelial neoplasia without evidence of prostate cancer)
* Patients on strong inhibitors of CYP1A2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Park, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (7):
- United States (7):
  - Seby B. Jones Cancer Center, Boone, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - Moses Cone Regional Cancer Center, Greensboro, North Carolina
  - Leo Jenkins Cancer Center, East Carolina University Medical Center, Greenville, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 patients were enrolled between March 2011 and May 2013.
Pre-assignment Details: 28 patients were assessed for eligibility; 4 patients were excluded for not meeting the inclusion criteria and 1 patient eventually declined to participate. Leaving 23 patients enrolled.
Period: Overall Study
Arm/Group | Bendamustine, Rituximab
Started | 23
Completed | 11
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 2
Not completed — Clinical deterioration | 1
Not completed — Physician Decision | 1
Not completed — Other complicating disease (stroke) | 1

BASELINE CHARACTERISTICS:
Groups:
- Bendamustine, Rituximab: This is a single arm intervention where patients will receive bendamustine at a dose of 120 mg/m^2 infused over 60 minutes in days 1 and 2 of each 21 day cycle along with rituximab 375 mg/m^2 after bendamustine on day 1 of each cycle. Patients with Eastern Cooperative Oncology Group (ECOG) PS of 3 at baseline were allowed to receive bendamustine at a dose of 90 mg/m^2 daily with a dose increase to 120 mg/m^2 daily if their ECOG improved.
  Bendamustine: Dosage Form: Intravenous (60 minute infusion) Dosage: 120mg/m2 (ECOG = 0-2) or 90mg/m2 (ECOG = 3) Frequency: Day 1 and Day 2; Every 3 weeks of a 21 day cycle. Duration: 3-6 Cycles
  Rituximab: Dosage form: Intravenous Dosage: 375 mg/m2 Frequency: Day 1 of every 3 weeks of a 21 day Cycle Duration: 3-6 Cycles
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 80 [65 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Stage [Count of Participants; unit: Participants] — stage I: 1 group of lymph nodes affected stage II: 2 or more groups of lymph nodes affected either above or below the diaphragm (muscle that separates the chest from the abdomen) stage III: lymph nodes affected on both sides of the diaphragm stage IV: lymphoma is found in organs outside the lymphatic system or in the bone marrow.
  Participants
    II | 4
    III | 7
    IV | 12
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status was developed by the Eastern Cooperative Oncology Group. It describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). 0 being fully active, able to carry on all pre-disease performance without restriction and 5 being dead.
  Participants
    0 | 2
    1 | 9
    2 | 6
    3 | 6
International Prognostic Index (IPI) [Count of Participants; unit: Participants] — International Prognosis Index is a clinical tool developed by oncologists to aid in predicting the prognosis of patients with aggressive non-Hodgkin's lymphoma. 0 points represent low-risk and higher numbers represent higher risk.
  Participants
    2 | 5
    3 | 5
    4 | 8
    5 | 5
Lactate Dehydrogenase (LDH) [Count of Participants; unit: Participants] — Lactate dehydrogenase (LDH) is an enzyme that helps the process of turning sugar into energy for your cells to use. It is often elevated in patients with lymphoma, but normal levels are associated with better response to therapy and longer survival.
  Participants
    Normal | 8
    Elevated | 15
Pathology Subtype [Count of Participants; unit: Participants] — Diffuse Large B-Cell Lymphoma (DLBCL) staging involves molecular classification into subtypes. Germinal Center has shown typically better survival than Non-Germinal Center
  Participants
    Non-Germinal Center | 12
    Germinal Center | 7
    Not Classified | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate as Defined by The International Harmonization Project for Response Criteria
Description: Complete response (CR) is defined as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. The complete response rate is the percentage of participants achieving a CR.
Time Frame: 2 years
Population: This represents the data after inclusion of the first 23 patients at the planned interim analysis. The data analysis was performed prior to the previously determined 3-year follow-up period because the study did not reach the initially planned sample size to determine the survival rates in a statistically significant manner as secondary objectives.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
percentage of participants | 52 [30.6 to 73.2]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR consists of the complete response rate + the partial response rate (percentage of participants achieving a complete or partial response). Complete response is defined by The International Harmonization Project for Response Criteria as the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Partial response is defined as regression of measurable disease and no new sites.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
percentage of participants | 78

3. Secondary Outcome: Partial Response Rate
Description: The percentage of participants achieving a partial response (PR). PR is defined by The International Harmonization Project for Response Criteria as regression of measurable disease and no new sites.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
percentage of participants | 26 [10.2 to 48.4]

4. Secondary Outcome: Estimate of Progression-Free Survival
Description: Progression-free survival (PFS) will be summarized using the Kaplan-Meier method. PFS was defined as the time from the start of treatment until lymphoma progression or death as a result of any cause. Progression was defined by The International Harmonization Project for Response Criteria as any new lesion or increase by ≥50% of previously involved sites from nadir.
Time Frame: 2 years with the median follow-up of 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
Months | 5.4 [3.8 to 10.2]

5. Secondary Outcome: Overall Survival
Description: This represents the Kaplan-Meier estimates of median overall survival defined as the time from start of treatment until death as a result of any cause.
Time Frame: 2 years with the median follow-up of 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
Months | 10.2 [3.8 to 13.3]

6. Secondary Outcome: Evaluate the Toxicity and Tolerability of Bendamustine in Combination With Rituximab
Description: The major grade 3 or higher adverse events were haematological toxicities. The results below include common haematological and non-haematological toxicities of grade 3 or higher. A complete record of all adverse events are reported in the adverse events section. National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0 were used to assess toxicity.
Time Frame: Adverse events were collected while patients were on active treatment. The median treatment time was 18 weeks.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Bendamustine, Rituximab
Number analyzed (Participants) | 23
percentage of patients
  Lymphopenia | 70
  Anemia | 26
  Neutropenia | 17
  Thrombocytopenia | 17
  Lymphocytosis | 4
  Fatigue | 13
  Anorexia | 9
  Hyperglycemia | 9
  Urinary Tract Infection | 9
  Arthralgia | 4
  Atrial Fibrillation | 4
  Cognitive Disturbance | 4
  Generalized Muscle Weakness | 4
  Heart Failure | 4
  Hypoalbuminemia | 4
  Hyponatremia | 4
  Infusion Related Reaction | 4
  Myalgia | 4
  Nausea | 4
  Pleural Effusion | 4
  Maculopapular Rash | 4
  Sepsis | 4
  Skin Infection | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on active treatment. The median treatment time was 18 weeks.
Arm/Group | Bendamustine, Rituximab
All-Cause Mortality (participants affected / at risk) | 17/23
Serious Adverse Events (participants affected / at risk) | 15/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine, Rituximab (N=23)
Anorexia (Metabolism and nutrition disorders) | 2
Death NOS (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Lung infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 2
Anemia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Creatinine increased (Investigations) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Gastric hemorrhage (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Stroke (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine, Rituximab (N=23)
Abdominal pain (Gastrointestinal disorders) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 13
Alkalosis (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 20
Anorexia (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 14
Atrial fibrillation (Cardiac disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 3
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac troponin I increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 10
Dehydration (Metabolism and nutrition disorders) | 4
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Edema face (General disorders) | 1
Edema limbs (General disorders) | 4
Ejection fraction decreased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 4
Fatigue (General disorders) | 20
Fever (General disorders) | 3
Flushing (Vascular disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypersomnia (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 19
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Hypotension (Vascular disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1 — Infection:viral
Infusion related reaction (General disorders) | 4
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 2
Lethargy (Nervous system disorders) | 1
Lip infection (Infections and infestations) | 1
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 17
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 — Elevated LDH
Mucosal infection (Infections and infestations) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — no description given
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — myoclonic spasms
Neutrophil count decreased (Investigations) | 10
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Restlessness (Psychiatric disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 6
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 14
Lymphocyte count increased (Investigations) | 1

LIMITATIONS AND CAVEATS:
The planned interim analysis was designed for futility (if ORR is less than 13/23 patients). It passed the futility criteria, but based on the survival rate at the time of interim analysis, the investigators decided to terminate the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days